CLINICAL TRIAL: NCT00988949
Title: Phase I, Randomized, Placebo Controlled Proof Of Mechanism Study To Determine Efficacy Of PF-04455242 In Blocking Spiradoline (PF-00345768) Stimulated Prolactin Release In Healthy Male Adult Subjects
Brief Title: Proof Of Mechanism Study To Determine Efficacy Of PF-04455242 In Blocking Spiradoline (PF-00345768) Stimulated Prolactin Release
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B1071004
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2010-01

CONDITIONS: Bipolar Depression
Keywords: Proof of mechanism study
MeSH Terms: conditions — Bipolar Disorder | interventions — 2-methyl-N-((2'-(pyrrolidin-1-ylsulfonyl)biphenyl-4-yl)methyl)propan-1-amine; spiradoline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PF-04455242 18 mg (Experimental): Subjects in this arm will receive a single 18 mg oral dose of PF-04455242 prior to spiradoline challenge
  Interventions: Drug: PF-04455242; Drug: spiradoline
- Placebo (Placebo Comparator): Subjects in this arm will receive placebo prior to spiradoline challenge.
  Interventions: Other: Placebo; Drug: spiradoline
- PF-04455242 30 mg (Experimental): Subjects in this arm will receive a single 30 mg oral dose of PF-04455242 prior to spiradoline challenge.
  Interventions: Drug: PF-04455242; Drug: spiradoline

INTERVENTIONS:
Drug: PF-04455242 — Single oral 18 mg dose of PF-04455242.
  Arms: PF-04455242 18 mg
Drug: spiradoline — Spiradoline 3.2 mcg/kg to be administered intramuscularly once on the morning of the spiradoline challenge day.
  Arms: PF-04455242 18 mg
Other: Placebo — Oral placebo.
  Arms: Placebo
Drug: spiradoline — Spiradoline 3.2 mcg/kg to be administered intramuscularly once on the morning of the spiradoline challenge day.
  Arms: Placebo
Drug: PF-04455242 — Single 30 mg oral dose of PF-04455242.
  Arms: PF-04455242 30 mg
Drug: spiradoline — Spiradoline 3.2 mcg/kg to be administered intramuscularly once on the morning of the spiradoline challenge day.
  Arms: PF-04455242 30 mg

SUMMARY:
This study will be a Proof of Mechanism (POM) study to establish evidence of central pharmacodynamic activity for PF 04455242, and will be a parallel group, randomized, double blind, sponsor open study conducted in healthy male subjects. Once subjects achieve steady state of PF 04455242, they will undergo PF 00345768 (spiradoline) challenge. Data will be analyzed to determine whether PF-04455242 blocks spiradoline induced prolactin release.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 21 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline area under the serum PRL concentration time curve from 0 to 120 minutes after intramuscular administration of PF 00345768 (spiradoline). | 1 week

SECONDARY OUTCOMES:
Change from baseline to peak of serum PRL concentration. | 1 week
Change from baseline to peak of plasma ACTH concentration. | 1 week
Change from baseline area under the plasma ACTH concentration time curve from 0-120 minutes after intramuscular administration of PF 00345768 (spiradoline). | 1 week
Plasma concentrations of PF 04455242. | 1 week
Clinical monitoring of safety and tolerability will include physical exam and neurological assessment, clinical safety laboratory results, 12 lead ECGs, vital signs, suicidality assessment, and adverse event monitoring | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1071004&StudyName=Proof%20Of%20Mechanism%20Study%20To%20Determine%20Efficacy%20Of%20PF-04455242%20In%20Blocking%20Spiradoline%20%28PF-00345768%29%20Stimulated%20Prolactin%20Release